CLINICAL TRIAL: NCT04001192
Title: Exercise in Patients With Post-Concussion Symptoms - a Pilot Study
Brief Title: Exercise in Patients With Post-Concussion Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018/2159
Record Dates: First submitted 2019-06-26; First posted 2019-06-27 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Craniocerebral Trauma; Head Injury, Minor; Postconcussion Syndrome; Posttraumatic Headache; Mild Traumatic Brain Injury
Keywords: exercise; exercise therapy; treadmill; symptom threshold; Postconcussion symptoms
MeSH Terms: conditions — Craniocerebral Trauma; Post-Concussion Syndrome; Post-Traumatic Headache; Brain Concussion; Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- exercise (Experimental): exercise at home, 5-6 days per week during 12 weeks, guided by a schedule that the physiotherapist will design after initial treadmill testing. Exercise intensity is 80-90 % of the heart rate threshold that was identified by the treadmill test. During the 12 weeks program, intensity will be increased according to feedback from the participant.
  Interventions: Behavioral: aerobic exercise program

INTERVENTIONS:
Behavioral: aerobic exercise program — The intervention is exercise at home, 5-6 days per week during 12 weeks, guided by a schedule that the physiotherapist will design after initial treadmill testing. Exercise intensity is 80-90 % of the heart rate threshold that was identified by the treadmill test. During the 12 weeks program, intensity will be increased according to feedback from the participant.

SUMMARY:
Physical activity and exercise have traditionally not been much of a focus in treatment of postconcussion symptoms and posttraumatic headache. On the contrary, patients have often got advice to rest until they were free from symptoms. This approach, however, is challenged, and complete rest should probably be discouraged after the first 24-72 hours. Moderate aerobic exercise has been found promising in the early phase after sports-related concussion, and in the treatment of patients with headache. This study is an open pilot-study of guided, home-based exercise in a clinical sample with postconcussion symptoms and posttraumatic headache after mixed-mechanism mild traumatic brain injury and minimal head injuries. The study will result in data about the feasibility and possible effects of exercise as treatment for prolonged postconcussion symptoms and posttraumatic headache.

ELIGIBILITY:
Inclusion Criteria:

* having sustained a minimal head injury (according to the Head Injury Severity Scale, HISS) or mild traumatic brain injury (TBI) (according to the TBI definition and the WHO criteria for mild TBI) within the last three years).
* post-concussion symptoms of at least moderate degree (according to the Rivermead postconcussion symptom questionnaire RPCSQ) occurring within the first week after the head injury and/or posttraumatic headache according to the International Classification of Headache Disorders 3 (ICHD-3) criteria.
* outpatients at St Olavs Hospital Clinic of Physical Medicine and Rehabilitation, Department of Acquired Brain Injury

Exclusion Criteria:

* Symptoms better explained by other conditions.
* Severe communication problems, typically due to language problems.
* Severe psychiatric, neurological, somatic or substance abuse disorders that will complicate follow-up and outcome assessment.
* Orthopedic injury or other disability too severe for performing the test or the intervention.
* Cardiovascular conditions or risk factors that are not compatible with testing or safe unsupervised exercise.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-02-14 (Actual); Primary Completion 2021-07-08 (Actual); Study Completion 2021-07-08 (Actual)

PRIMARY OUTCOMES:
The proportion of participants completing the exercise program | 12 weeks
Estimated change in post concussion symptom burden | 12 weeks
  assessed with Rivermead postconcussion symptom questionnaire (www.tbi-impact.org/cde/mod_templates/12_F_06_Rivermead.pdf) 17 questions about severeness of symptoms, answers 0 (not experienced at all) - 4 (a severe problem). Ratings on the total symptom scores, and for individual items..

SECONDARY OUTCOMES:
Change in posttraumatic headache | 12 weeks
  Change in number of days with moderate or severe headache during the last 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bjørn Skogstad, md, Study Director — St. Olavs Hospital; Toril Skandsen, md phd, Principal Investigator — St. Olavs Hospital
Locations (1):
- St Olavs Hospital, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No